CLINICAL TRIAL: NCT03959605
Title: Genetic Determinant of Foveolar Hypoplasia in Parents of Albinos Children
Acronym: ALAFOR
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: MMT_2019_2
Record Dates: First submitted 2019-05-18; First posted 2019-05-22 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Albinism, Ocular
MeSH Terms: conditions — Albinism, Ocular | interventions — Blood Specimen Collection; Genetic Testing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: blood sample for genetic test — detection of pathogenic variants among the 19 genes known to be involved in albinism
Diagnostic Test: Ophtalmological examination — measurement of visual acuity, OCT and OCTA

SUMMARY:
Fovea plana could be the phenoyipic translation of a genetic anomaly in one of the genes identified in albinisme

ELIGIBILITY:
Inclusion Criteria:

* children with albinism
* father and mother of children with albinism

Exclusion Criteria:

* sign of albinism except fovea plana in father or mother of children with albinism
* ophthalmological abnormalities making access to the fundus with OCT impossible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: parents without symptom of albinism (except fovea plana) of children with albinism
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2019-01-06 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Number of genetics variants | 1 month
  among the genes involved in albinism, identification of those presents in parents of children with albinism

CONTACTS AND LOCATIONS:
Overall Officials: Martine MAUGET FAYSSE, Principal Investigator — Fondation A. de Rothschild
Locations (1):
- Fondation A de Rothschild, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided